CLINICAL TRIAL: NCT06916364
Title: Utilization of Airway Stabilizing Rod to Assist With Laryngeal Mask Airway Guided Fiberoptic Intubation in Adults With Obesity
Acronym: FASTER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kevin W Duong, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-55523
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Adult; Obesity, Morbid
Keywords: faster; Laryngeal mask airway guided intubation; Fiberoptic Intubation; Airway Stabilizing Rod
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Morbid Obesity (Experimental): Elective surgery requiring intubation, Age > 18, BMI > 35 kg/m2
  Interventions: Device: Fiberoptic Assisted Endotracheal Rod Intubation

INTERVENTIONS:
Device: Fiberoptic Assisted Endotracheal Rod Intubation — Fiberoptic-Assisted Endotracheal Rod for Endotracheal Intubation Through a Supraglottic Airway
  Other Names: FASTER

SUMMARY:
The FASTER stabilizing rod offers the distinct advantage of intubating through the laryngeal mask airway with a fiberoptic scope via the FASTER stabilizing rod. The device allows for the provider to insert the endotracheal tube (ETT) with visual confirmation using the fiberoptic scope into the trachea. The device then allows for the laryngeal mask airway to be removed while stabilizing the ETT to ensure the ETT does not get dislodged.

The purpose of this protocol is to clinically test the validated prototype that the investigators have built and previously tested in adults with obesity.

The primary aims are to evaluate 1) the time to intubation and 2) the number of intubation attempts. The secondary aim is to note any complications from time to intubation to PACU discharge.

These complications include: Hypoxemia (10% decrease from baseline for 45 seconds)1 Airway trauma (minor) Esophageal intubation Laryngospasm Bronchospasm Oro-pharyngeal bleeding Arrythmia Emesis Epistaxis Dental damage Post-operative sore throat Post-operative hoarseness Accidental extubation during removal of the LMA.

DETAILED DESCRIPTION:
When a patient cannot be ventilated and/or intubated, the guidelines for airway management (ASA difficult airway algorithm) dictate that a laryngeal mask airway (LMA) be used as a rescue device to oxygenate and ventilate the patient. However, an LMA is generally temporary and ultimately needs to be replaced by an endotracheal tube (ETT).

At present, providers can use an exchange catheter through the LMA to place the ETT. However, all current techniques to place the ETT through the LMA are done WITHOUT direct visualization or the ability to provide oxygenation or ventilation. This has the possibility of either accidental tracheal extubation or esophageal intubation as well as the possibility of causing trauma to the airway, particularly of concern in a patient with a difficulty airway.

To bridge this gap, the investigators developed an innovative device called the FASTER that would allow for patients (children through adults) to have an ETT placed through the LMA under direct vision and while being able to oxygenate and ventilate, greatly improving safety.

The first step was to create a prototype that was validated in a mannequin (H-47253 ). Following this validation, the investigators created and successfully performed a feasibility study in children without difficult airway at Texas Children's demonstrating success and no adverse events (H-47253) . Following this feasibility study, and despite the FASTER device being completely external to the patient, given that the study was performed in children, the investigators obtained an IDE from the FDA for study in children specifically with difficulty airways. At present, the investigators have successfully completed an initial study in children (n=20) (H-50120) all with difficulty airways without any adverse events. In this study, children that were previously difficult to intubate having an average of three intubating attempts were intubated in a single attempt in an average of just 66 seconds.

The objective for this protocol is to demonstrate feasibility in using this device in adult obese patients. In this study, the investigators will be using this device that is completely external to the patient and only in adults (not including any protected classes of patients).

Moreover, in the completed study of children with actual difficulty airways, the investigators demonstrated tremendous success and patient benefit without any adverse events. In this protocol, the investigators will not enroll any patients with difficult airway nor any patients in protected classes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-64 yrs),
* Geriatric (65+ yrs)
* BMI > 35 kg/m2
* elective surgery requiring intubation

Exclusion Criteria:

* pregnant woman
* neonates
* children
* incarcerated patient
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to Intubation | 3 minutes
  Time of disconnecting the circuit from supraglottic airway (SGA) to the presence of end tidal carbon dioxide (ETCO2) for intubation.
Number of Intubation Attempts | 5 minutes
  Defined as failure to capture end tidal carbon dioxide after completion of intubation.

SECONDARY OUTCOMES:
Complications | Up to 1 day
  These complications include number of participants with
  * Hypoxemia (10% decrease from baseline for 45 seconds)
  * Airway trauma (minor)
  * Esophageal intubation
  * Laryngospasm
  * Bronchospasm
  * Oro-pharyngeal bleeding
  * Arrhythmia
  * Emesis
  * Epistaxis
  * Dental damage
  * Post-operative sore throat
  * Post-operative hoarseness
  * Accidental extubation during removal of the LMA

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kovatsis PG. Continuous ventilation during flexible fiberscopic-assisted intubation via supraglottic airways. Paediatr Anaesth. 2016 Apr;26(4):457-8. doi: 10.1111/pan.12863. No abstract available. PMID 26956516
- [Background] van Zundert TC, Wong DT, van Zundert AA. The LMA-Supreme as an intubation conduit in patients with known difficult airways: a prospective evaluation study. Acta Anaesthesiol Scand. 2013 Jan;57(1):77-81. doi: 10.1111/aas.12011. Epub 2012 Nov 21. PMID 23167262
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Joffe AM, Aziz MF, Posner KL, Duggan LV, Mincer SL, Domino KB. Management of Difficult Tracheal Intubation: A Closed Claims Analysis. Anesthesiology. 2019 Oct;131(4):818-829. doi: 10.1097/ALN.0000000000002815. PMID 31584884